CLINICAL TRIAL: NCT05316623
Title: Using Peripheral Neurostimulation to Improve Work Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Collaborators: Réseau Provincial De Recherche En Adaptation-Réadaptation (REPAR) (Unknown); Réseau québécois de recherche sur le vieillissement (RQRV) (Unknown)
Responsible Party: Principal Investigator, Guillaume Léonard, Professor, Université de Sherbrooke
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: 2019-2885
Record Dates: First submitted 2022-03-15; First posted 2022-04-07 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: One placebo group and one intervention group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Sham Comparator): Simulated TENS and personalized exercise program in telerehabilitation (3 sessions/week over 3 weeks) n = 12
  Interventions: Device: TENS
- Intervention group (Experimental): Real TENS and personalized exercise program in telerehabilitation (3 sessions/week over 3 weeks) n = 12
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — TENS (strong and comfortable intensity) applied during exercises in a telerehabilitation setting.
  Other Names: Transcutaneous electrical nerve stimulation; Peripheral neurostimulation

SUMMARY:
Physical exercise plays a central role in work rehabilitation. However, the presence of pain (particularly common in older adults and aging workers) can lead to a fear of movement (kinesiophobia) and hinder rehabilitation. Access to rehabilitation care is also a barrier for many older adults, which could be circumvented through telerehabilitation. The objective of this pilot study is to document the feasibility and explore the effect of a telerehabilitation intervention combining therapeutic exercises and real TENS (experimental group) or placebo TENS (control group) in individuals aged 55 and over who have stopped working (triple-blind randomized controlled study). To do so, various feasibility indicators (e.g., recruitment rate, adherence) and clinical measures (e.g., kinesiophobia, pain during exercise) will be documented before and after the intervention. Together, these measures will help assess the appropriateness of conducting a large-scale study aimed at potentiating work rehabilitation in older populations.

DETAILED DESCRIPTION:
Problem and hypotheses:

In 2019, the proportion of Canadians aged 55 and over who were employed was 35.9%, the highest rate recorded to date since 1976. Despite their willingness to remain employed, seniors are more prone to work disability and early retirement. Older workers with disabilities are particularly vulnerable to job retention. In Quebec, the average length of absence following a work-related injury is 134 days for workers aged 55 and over, while it is less than 50 days for those aged 15 to 24. This difference can be explained in part by the presence of persistent pain that disproportionately affects older individuals and can significantly impede rehabilitation to work. The indirect costs associated with unemployment and absenteeism of people living with chronic pain were estimated to be $22.5 billion in Canada in 2019. A recent review conducted and published by our team found that strategies to reduce pain are one of the most important elements to consider in enabling workers to remain in the workplace after an episode of musculoskeletal disorder.

Exercise plays a central role in chronic pain management and work rehabilitation. However, pain can be a major barrier to physical activity. Therefore, finding ways to reduce pain during and after exercise is essential to facilitate rehabilitation. Peripheral neurostimulation (TENS) - an electrotherapeutic modality that uses an electrical current to depolarize peripheral nerve fibers with electrodes applied directly to the skin - is effective in temporarily relieving pain. It represents an interesting avenue for increasing exercise tolerance associated with exercise in the pain subject. To date, 3 studies have investigated the use of TENS during exercise, all showing positive results. None, however, have yet investigated this strategy (TENS + exercise) in aging workers living with persistent pain.

We postulate that telerehabilitation treatments (therapeutic exercises) provided concurrently with actual TENS will be more effective in reducing the biopsychological impacts of pain than the same rehabilitation treatments paired with placebo TENS. Thus, our hypothesis is that the experimental treatment will cause participants to enter a "virtuous circle": the TENS will allow for a punctual reduction of pain and kinesiophobia, which will encourage the realization/resumption of activity and lead to sustained benefits (e.g., physical function, pain, mood).

Objectives:

The primary objective of this pilot study is to explore the feasibility and acceptability of using real TENS, compared to placebo TENS, as a complementary treatment to a telerehabilitation exercise program, in workers who are off work.

The secondary objective is to compare the effect of the two types of intervention (real TENS + exercises vs. placebo TENS + exercises) on clinical outcomes (e.g. pain intensity, functioning in vocational rehabilitation, etc.).

Methods and analysis:

Design:

This project consists of a randomized controlled trial following a quadruple blind design.

Participants:

The target population is aging workers who are off work due to a musculoskeletal injury.

Sampling and recruitment procedures:

Participants will be recruited at the ISO-SANTÉ and Physio-Atlas clinics in Sherbrooke, which specialize in work rehabilitation (volunteer, non-probability sampling). The recruitment of individuals will be done through posters and with the help of clinicians who will be invited to talk to patients about the project.

Conduct of the study:

The purpose of this study is to recruit 24 participants who will take part in an exercise program spread over 3 weeks, with 3 sessions per week. The duration of each session is 30 minutes. The exercise program will be determined by the research team, in collaboration with clinic health professionals, and the exercises will be delivered via the TeraPlus telerehabilitation platform. The TENS (real or simulated) will be worn by participants throughout their telerehabilitation exercises, under the supervision of the student researcher.

ELIGIBILITY:
Inclusion Criteria:

* Being 55 years of age or older
* Being off work completely due to a musculoskeletal injury
* Starting a physical rehabilitation program
* Being in employment
* Experiencing pain of mild intensity (score of 1-3 points on a numerical scale of 0-10 points) to moderate intensity (score of 4-6 points) during movements/exercises
* Being comfortable enough with technology to participate in video conferences, respond to emails or text messages
* Having stable medication and lifestyle habits
* Speaking French

Exclusion Criteria:

* Having a cognitive deficiency
* Wearing a cardiac defibrillator or pacemaker
* Being diagnosed with cancer
* Having already experimented with TENS

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 4 months
  The number of participants randomized divided by the number of participants screened.
Exclusion rate | 4 months
  The number of ineligible participants divided by the number of participants screened.
Refusal rate | 4 months
  The number of participants who refused to participate in the trial divided by the number of participants screened.
Adherence rate | 3 weeks
  The number of people who finished intervention divided by the number of participants randomized.
Attrition rate | 3 weeks
  The number of people who did not finish intervention divided by the number of participants randomized.
Kinesiophobia | 3 weeks
  excessive, irrational, and debilitating fear of physical movement and activity resulting from a feeling of vulnerability due to painful injury or reinjury - Measured with the Tampa scale of kinesiophobia

SECONDARY OUTCOMES:
Severity of pain and impact of pain on physical function | 3 weeks
  Measured with the Brief Pain Inventory (BPI)
Pain intensity | 3 weeks
  Measured with a visual analog scale (VAS). Scale from 0 to 100, where 0 indicates no pain and 100 indicates worst pain imaginable
Psychosocial component and impact of pain on the emotional sphere | 3 weeks
  Measured with Beck's depression inventory. Contains 21 items with a 4-point likert scale. The minimum possible score is 0 and the maximum possible score is 63. The higher the score, the more important the psychosocial component is for the individual.
Qualitative component of pain | Intervention period (before first and after last sessions)
  McGill Pain Questionnaire (MPQ). The MPQ is composed of 20 questions and scores range from 0 (no pain) to 78 (severe pain).
Pain catastrophizing | 3 weeks
  Measured with the Pain Catastrophizing Scale. It consists of 13 thoughts or emotions related to a painful experience. Each thought is scored on 5 points from 0 to 4. The total score is 52 points. If the score is between 20 and 29, the risk of pain chronicization is moderate. If the score is between 29 and 52, the risk is high. The higher the score, the higher the risk.
Disability in work Rehabilitation | 3 weeks
  Measured with the Work Rehabilitation Questionnaire (WORQ). The WORQ is used to better understand the extent of problems in functioning that people may have due to their health condition(s) and who are undergoing work or vocational rehabilitation. In the main section, responders rate the extent of their problem in the past week on a scale from 0 (no problem) to 10 (complete problem / not possible).
Overall treatment satisfaction | 3 weeks
  Measured with The self-report measure Patient Global Impression of Change (PGIC). PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Quality of movement | 3 weeks
  Measuring the posture of the participants during the execution of a squat (sagittal view on camera). Based on the Back Squat Assessment.
Quality of movement | 3 weeks
  Measuring the posture of the participants during the execution of a squat (sagittal view on camera). Based on the squat portion of the New Basic Functional Assessment Protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Léonard, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche sur le vieillissement (CdRV), Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No